CLINICAL TRIAL: NCT00857675
Title: A Multi-Centre, Double-Blind , Randomized, Placebo-Controlled Phase II/III Study of Adefovir Dipivoxil for the Treatment of Chinese Patients With HBeAg Positive Chronic Hepatitis B Followed by Long-Term (5 Years Total) Adefovir Dipivoxil Treatment. (Report on Year 1 and Year 2 Data)
Brief Title: A Efficacy and Safety Study of Adefovir Dipivoxil to Treat Chinese Patients With HBeAg+ve Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADF30001
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Hepatitis B
Keywords: HBV DNA suppression; ALT normalisation; Viral resistance; HBeAg seroconversion
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Adefovir Dipivoxil (Experimental): ADV 10mg tablets once daily
  Interventions: Drug: AAAA; Drug: AAPA; Drug: PAAA
- Adefovir Dipivoxil matched placebo (Placebo Comparator): Adefovir Dipivoxil matched placebo one tablet once daily
  Interventions: Drug: AAPA; Drug: PAAA

INTERVENTIONS:
Drug: AAAA — Adefovir Dipivoxil (12 weeks) + open lable Adefovir Dipivoxil (28 weeks) + Adefovir Dipivoxil (12 weeks) + Open label Adefovir Dipivoxil (52-260weeks)
  Arms: Adefovir Dipivoxil
Drug: AAPA — Adefovir Dipivoxil (12 weeks) + Open label Adefovir Dipivoxil (28 weeks) + placebo (12 weeks) + open label-Adefovir Dipivoxil (52-260 weeks)
Drug: PAAA — Placebo (12 weeks) + Open label Adefovir Dipivoxil (28 weeks) + Adefovir Dipivoxil (12 weeks) + Open label Adefovir Dipivoxil (52-260 weeks)

SUMMARY:
The purpose of this study is to determine whether Adefovir Dipivoxil is effective and safe in treatment of Chinese Patients with HBeAg positive Chronic Hepatitis B for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Presence of HBsAg and HBeAg at the time of screening and for at least 6 months prior to screening.
* Positive HBV DNA plasma assay with screening value equal or more than 10 (6) copies/mL (Roche COBAS AMPLICORTM HBV MONITOR Test, LLOD less than 300 copies/mL) at the time of screening (within 4 weeks of randomisation).
* Evidence of elevated serum ALT levels defined as serum ALT level greater than or equal to 2.0 times (inclusive) the upper limit of the normal range (ULN) in the previous 6 months, and serum ALT levels greater than 1.0 times the ULN at the time of screening.

Exclusion Criteria:

* Evidence of hepatocellular carcinoma;
* Clinical signs of liver decompensation;
* Serum creatinine more than 1.5 mg/dL;
* ALT more than 10 x ULN; seropositivity for hepatitis C or D virus or HIV;
* Lamivudine therapy within 3 months prior to screening;
* ADV therapy or any other anti-HBV therapy within the previous 6 months;
* Use of systemic antiviral agents, immunomodulators, immunosuppressive therapy, Chinese Traditional Medicines or agents known to lower ALT levels during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2002-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The log10 reduction in HBV DNA from baseline at week 12 between ADV 10mg and matching placebo | Week 12

SECONDARY OUTCOMES:
The proportion of subjects with ALT normalisation | Week 52, 104, 156, 208, 260
log10 reduction in serum HBV DNA | Week 52, 104, 156, 208, 260
The proportion of subjects with HBV DNA 10(5) copies/mL or a 2 log10 reduction from Baseline HBV DNA level | Week 52, 104, 156, 208, 260
The proportion of subjects with HBeAg loss | Week 52, 104, 156, 208, 260
The proportion of subjects with HBeAg seroconversion | Week 52, 104, 156, 208, 260
The proportion of subjects developing N236T and A181V HBV DNA genotypic mutations associated with ADV resistance | Week 52, 104, 156, 208, 260
The proportion of subjects with HBV DNA undetectable (<300 copies/mL) | Week 52, 104, 156, 208, 260

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- China (8):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Chongquin
  - GSK Investigational Site, Shanghai